CLINICAL TRIAL: NCT06719414
Title: A Multi-center Study on Amide Proton Transfer-Weighted Imaging in Predicting Pathological Complete Response After Neoadjuvant Therapy of Rectal Cancer
Brief Title: Application of Amide Proton Transfer-Weighted Imaging in Predicting Pathological Complete Response After Neoadjuvant Therapy of Rectal Cancer
Status: Recruiting | Type: Observational
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Collaborators: Xinyi People's Hospital (Unknown)
Responsible Party: Principal Investigator, Peiyi Xie, associate chief physician, Sixth Affiliated Hospital, Sun Yat-sen University
Other Study IDs: 2024ZSLYEC-552
Record Dates: First submitted 2024-11-27; First posted 2024-12-05 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to learn about the amide proton transfer-weighted imaging for rectal cancer response assessment after neoadjuvant therapy. The main question it aims to answer is:

• Does amide proton transfer-weighted imaging predict the cancer response before surgery? Participants will underwent amide proton transfer-weighted imaging as part of their regular MRI examination.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced rectal cancer(cT3-4, or cN+), resectable, histologically confirmed rectal adenocarcinoma
* Received neoadjuvant therapy before surgery
* Complete radical resection of rectal cancer and postoperative pathological examination
* Informed consent and signed the informed consent form

Exclusion Criteria:

* Poor image quality, such as severe artifacts
* Complicated with intestinal obstruction, intestinal perforation and other cases requiring surgical treatment
* The interval between preoperative MRI and surgery was more than 2 weeks
* Prior treatment for rectal cancer
* History of other malignant tumors
* Patients who cannot undergo MRI examination due to contraindications or relative contraindications
* Patients were lost to follow-up or voluntarily withdrew from the study due to adverse reactions or other reasons

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally advanced rectal cancer treated with neoadjuvant therapy
Sampling Method: Non-Probability Sample
Enrollment: 320 (Estimated)
Dates: Start 2024-10-22 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
the area under curve (AUC) of receiver operating characteristic (ROC) curves of models in prediction tumor response | From date of baseline MRI to date of preoperative MRI，within 12 months

SECONDARY OUTCOMES:
the specificity of models in prediction tumor response | From date of baseline MRI to date of preoperative MRI，within 12 months
the sensitivity of models in prediction tumor response | From date of baseline MRI to date of preoperative MRI，within 12 months
the positive predictive value of models in prediction tumor response | From date of baseline MRI to date of preoperative MRI，within 12 months
the negative predictive value of models in prediction tumor response | From date of baseline MRI to date of preoperative MRI，within 12 months
the accuracy of models in prediction tumor response | From date of baseline MRI to date of preoperative MRI，within 12 months
disease-free survival and overall survival | From date of enrollement until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sixth Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Xinyi People's Hospital, Maoming, Guangdong

IPD SHARING:
Plan to Share IPD: No